CLINICAL TRIAL: NCT03280342
Title: Cognitive Effects of Immediate Release Topiramate vs Extended Release Topiramate in Patients With Migraine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study
Sponsor: University of Minnesota (Other)
Collaborators: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FWA00000312-10
Record Dates: First submitted 2017-09-01; First posted 2017-09-12 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Migraine; Headache
Keywords: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Topiramate

STUDY DESIGN:
Intervention Model Description: a crossover, randomized, double blind design in conjunction with intensive pharmacokinetic sampling and multiple administrations of a neurocognitive test battery to directly compare the effects on cognition of IR-TPM to XR-TPM in adults with migraine. The dose will begin at 25mg and titrated in 25mg increments to reach target dose of 100mg.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IR-TPM (Topamax) (Active Comparator): IR-TPM (Topamax)
  Interventions: Drug: IR-TPM (Topamax); Drug: XR-TPM (Trokendi XR)
- XR-TPM (Trokendi XR) (Active Comparator)
  Interventions: Drug: IR-TPM (Topamax); Drug: XR-TPM (Trokendi XR)

INTERVENTIONS:
Drug: IR-TPM (Topamax) — XR-TPM (Trokendi XR)
Drug: XR-TPM (Trokendi XR) — XR-TPM (Trokendi XR)

SUMMARY:
Crossover, randomized, double blind: Q12h dosing in both periods; matching placebo for evening dosing during XR treatment; target dose: 100mg

DETAILED DESCRIPTION:
The primary objective is to compare the effect of treatment with an immediate-release topiramate (IR-TPM), namely Topamax®, to an extended-release topiramate (XR-TPM), namely Trokendi XR®, regimen on cognition in adults with migraine.

The secondary objective is to determine the factors that explain inter-individual variability in cognitive response. Pharmacokinetic and demographic factors will be explored. Variability in cognitive response between individuals can be large. A population approach (nonlinear, mixed effects) will be used to determine drug exposure response relationships.

ELIGIBILITY:
Inclusion Criteria:

1. Established history of episodic migraine with or without aura, as assessed by International Headache Society criteria, for at least 6 months before screening and frequency of 3 or more headache attacks per month during the past 3 months
2. Male or female, ages 18-65
3. Women are required to be postmenopausal, surgically incapable of bearing children, or practicing a medically acceptable method of birth control (i.e., double barrier method, IUD, Mirena, etc) for at least 1 month before study entry through 30 days following last dose.
4. If postmenopausal and on hormone replacement therapy (HRT) then must to be on a stable regimen for at least 2 months (continuous stable regimen of cyclic or non-cyclic HRT); negative pregnancy test.
5. Native English speakers (due to speech and language analysis)
6. Montreal Cognitive Assessment (MoCA) score equal to or greater than 26.

Exclusion Criteria:

1. Onset of migraine occurred after age 50 years, or overuse of analgesics or migraine specific agents for the acute treatment of migraine episodes; examples of analgesic overuse included the following: more than 8 treatment episodes (episode defined as any calendar day of usage) of ergot containing medications a month; more than 8 treatment episodes of triptans a month; or more than 6 treatment episodes of potent opioids a month.
2. Required, continued use of the following medications for any medical reason during the study: beta-blockers, benzodiazepines, tricyclic antidepressants, antiepileptics, calcium channel blockers, monoamine oxidase inhibitors, nonsteroidal anti-inflammatory drugs (NSAIDs) daily, opioids, agents for insomnia (e.g., Ambien, diphenhydramine-containing OTC products); corticosteroids, local anesthetics, botulinum toxin within last three months, or herbal preparations such as feverfew or St John's wort. However, subjects will be permitted to be on a stable regimen of a selective serotonin reuptake inhibitor or SNRI for 3 months or more for depression and/or anxiety.
3. A history of nephrolithiasis
4. Have previously taken topiramate
5. Received an experimental drug or used an experimental or approved device for migraine prevention (e.g., TENIS unit) within 30 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Controlled Oral Word Association Test (COWA)-generative phonemic fluency | Baseline (Day 1) through Day 52
  The primary outcome measure is the Controlled Oral Word Association (COWA: phonemic generative fluency). COWA was chosen as the primary endpoint since in previous studies of drug-induced cognitive impairment, this measure was sensitive to the effects of topiramate (Meador et al, 2003; Marino et al, 2012; Marino et al, 2015). The primary endpoint is a change in the COWA score from baseline to each post-dose assessment

SECONDARY OUTCOMES:
Measures of semantic verbal fluency | Baseline (Day 1) through Day 52
  Change in scores from individual baseline to each post-dose assessment on measures of semantic verbal fluency (e.g., Animals)
Digit Span Backward | Baseline (Day 1) through Day 52
  Change in scores from individual baseline to each post-dose assessment on measures of working memory (i.e., Digit Span Backward)
Digit Symbol Modalities Test (SDMT) | Baseline (Day 1) through Day 52
  Change in scores from individual baseline to each post-dose assessment on measure of psychomotor speed
Trails A & B | Baseline (Day 1) through Day 52
  Change in scores from individual baseline to each post-dose assessment on measures of executive function

CONTACTS AND LOCATIONS:
Overall Officials: Susan Marino, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Prism Research, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No